CLINICAL TRIAL: NCT06918197
Title: Evaluation the Impact of the "Pas" Technique Versus the "Standard" Technique on Radiation Exposure, Procedure Efficiency, and Patient Outcome in Pain Management Injections
Brief Title: Evaluation the Impact of the "Pas" Technique Versus the "Standard" Technique on Radiation Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthospine Advance Health, Inc. (Other)
Responsible Party: Principal Investigator, Gabriel Garcia-Diaz, Orthopedic Spinal Surgeon, Principal Investigator, Mercy Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#2023-099
Record Dates: First submitted 2024-11-03; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Spine; Fluoroscopy for Spine Surgery; Back Pain; Sacroiliac Joint
Keywords: Spine; PAS
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Technique (Active Comparator): Standard Technique is the standard protocol for the pain management procedures completed in this study such as Medical Branch Block, Radiofrequency Ablation, Sacroiliac Joint Block, and Transforaminal Epidural
  Interventions: Procedure: Standard Technique
- PAS Technique (Experimental): PAS Technique Protocol:
  The following steps outline the PAS Technique. While the example below uses 6 injection sites, the approach can be adapted for different pain management procedures with a different number of needle injection sites as needed.
  Timer: Begin stopwatch for entire procedure from start to medication insertion. Positioning: The patient is placed in a prone position on the fluoroscopic table. Time out was performed.
  Skin Preparation: Clean the injection site with an antiseptic solution and drape it to maintain sterility.
  Anesthesia: Administer intravenous sedation Identification of Anatomical Landmark:The spinous process was located and marked as the reference point (SP), which was then used as a guide for the following steps.
  Marking Target Points: Using the spinous process (SP) as the anatomical landmark and X-ray guided fluoroscopy, Target Point 1 (TP1) was identified and its position verified. The X value (the horizontal distance from the SP to TP1) was measured.
  Interventions: Procedure: PAS Technique

INTERVENTIONS:
Procedure: PAS Technique — PAS Technique Protocol:
  The following steps outline the PAS Technique. While the example below uses 6 injection sites, the approach can be adapted for different pain management procedures with a different number of needle injection sites as needed.
  Timer: Begin stopwatch for entire procedure from start to medication insertion. Positioning: The patient is placed in a prone position on the fluoroscopic table. Time out was performed.
  Skin Preparation: Clean the injection site with an antiseptic solution and drape it to maintain sterility.
  Anesthesia: Administer intravenous sedation Identification of Anatomical Landmark:The spinous process was located and marked as the reference point (SP), which was then used as a guide for the following steps.
  Marking Target Points: Using the spinous process (SP) as the anatomical landmark and X-ray guided fluoroscopy, Target Point 1 (TP1) was identified and its position verified. The X value (the horizontal distance from the SP to TP1) was measured.
  Arms: PAS Technique
Procedure: Standard Technique — In the "Standard" or "Traditional "technique, the spinal needles are used to localize the anatomical objective using fluoroscopic guidance for each needle placement. Traditionally, each needle is placed individually with a spot radiological view before placement and after placement of each needle to confirm the localization.
  Arms: Standard Technique

SUMMARY:
The purpose of this study is to compare both techniques and analyze the data from the "Standard" technique to help design the "PAS" technique. In the "PAS" technique, investigators predetermine the distances from the needles and place them all together using our initial target needle marker in the objective anatomic landmark. Will randomized patients assigning them either in cohort 1 control "Standard" of care technique and cohort 2 "PAS" technique. After only utilizing the "Standard" of care technique, will obtain the measurements and distances from the needles inserted in patients under fluoroscopic guidance for the different pain procedures. The data will help demonstrate that is possible to predict the needle placement replicating with confidence good outcomes using the "PAS" technique to reduce the radiation exposure and time. Our data will justify the use of the "PAS" technique to become an alternative to the "Standard" of care technique for a faster, efficient, and replicable needle placement for diminished radiation exposure, to avoid complications and consistent good outcomes

DETAILED DESCRIPTION:
PAS Technique Protocol:

The following steps outline the PAS Technique. While the example below uses 6 injection sites, the approach can be adapted for different pain management procedures with a different number of needle injection sites as needed.

Timer: Begin stopwatch for entire procedure from start to medication insertion. Positioning: The patient is placed in a prone position on the fluoroscopic table. Time out was performed.

Skin Preparation: Clean the injection site with an antiseptic solution and drape it to maintain sterility.

Anesthesia: Administer intravenous sedation Identification of Anatomical Landmark:The spinous process was located and marked as the reference point (SP), which was then used as a guide for the following steps.

Marking Target Points: Using the spinous process (SP) as the anatomical landmark and X-ray guided fluoroscopy, Target Point 1 (TP1) was identified and its position verified. The X value (the horizontal distance from the SP to TP1) was measured. This X value was not just a guide but the exact horizontal distance used for the placement of all subsequent target points. For the vertical distance between target points, a consistent distance of 3 cm was applied. This value was determined as the average vertical distance between the target points based on prior findings.

Refer to Figure 2 for a detailed illustration of the target point positions in relation to the spinous process and the distances applied.

Horizontal Distance (X Values):

The X value represents the horizontal distance from the spinous process (SP) to each target point (TP).

The X value measured for TP1 was used as the fixed horizontal distance for all target points on both sides of the SP.

For target points on the opposite side of the SP, the same X value was mirrored.

Thus, for the entire procedure:

TP1 and TP4 were placed at an equal X distance to the right and left of the SP, respectively.

TP2 and TP5 followed the same X distance as TP1 and TP4, located on their respective sides of the SP.

Vertical Distance (Y Values):

The Y value represents the vertical distance between the target points. A consistent vertical distance was applied between the target points. This was determined as the average distance between the target points based on prior findings.

Therefore:

TP2 was positioned 3 cm below TP1. TP3 was positioned 3 cm above TP1. TP5 was positioned 3 cm below TP4. TP6 was positioned 3 cm above TP4.

Final Verification: One final fluoroscopic image was taken to verify the accurate placement of all needles at the marked target points.

ELIGIBILITY:
**Inclusion Criteria:**

* Adult patients aged 19 and older
* No history of:
* Convictions
* Infections
* Cancer
* Contraindications for surgical procedures
* Patients scheduled for pain injections who:
* Agree to participate in the study
* Sign informed consent and IRB approval consent
* Complete preoperative, postoperative, and 1-week postoperative questionnaires
* Patients with chronic lower back pain (lasting over three months) that has not responded to conventional treatments (e.g., NSAIDs, back muscle strengthening, physiotherapy)
* Symptoms indicating facet pain, including:
* Lower back pain with or without radiation to the buttocks, thigh, or groin
* Pain increasing on hyperextension
* Pain during initial movements
* Focal tenderness over the facet joint when pressed
* Post-lumbar disc surgery patients with persistent pain but no MRI evidence of arachnoiditis or infection
* All procedures conducted under fluoroscopic guidance for spinal needle placement
* Data collection parameters:
* Gender, race, height, weight, BMI
* Radiation exposure from fluoroscopy dosage logbook
* Procedure time
* Horizontal and longitudinal distance measurements between spinal levels (in cm)
* Study period: October 1, 2023, to May 15, 2024

**Exclusion Criteria:**

* Evidence of:
* Infection (elevated WBC >12,000 or UTI)
* Neoplastic disease
* Possible pregnancy, bleeding diathesis, or anticoagulant therapy
* History of sensitivity to local anesthetics

**Preoperative and Postoperative Assessments:**

* Visual Analog Scale (VAS)
* Numeric Pain Scale
* Disability Oswestry Index questionnaires
* Additional data collection for both cohorts:
* Patient demographics (age, gender, race, height, weight, BMI)
* Radiation exposure from fluoroscopy (in mGy)
* Procedure duration
* Horizontal and vertical distance measurements (in cm) between spinal needle placements

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Radiation Exposure | through study completion, an average of 6 months
  Examined Radiation Exposure amount from Fluoroscopic Guidance on Patient
Radiation Exposure | During the index procedure (from first fluoroscopy activation to last activation on Day 0; ≤ 20 min)
  radiation exposure from the fluoroscopy dosage logbook
Procedure length in time | During the index procedure (from anesthesia induction to application of the final bandage after injection on Day 0; measured in minutes)
  Total Procedure Time

SECONDARY OUTCOMES:
Numeric Pain Scale | through study completion, an average of 6 months
  Examined Pain Index's before and After procedure
  Numeric Pain Scale from 1-10, one being the least pain and ten being the most- higher the pain score, the worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Oster, Metrowest IRB Chair, Study Chair — Metro West Medical Center
Locations (1):
- University Surgery Center, Merced, California, United States

IPD SHARING:
Plan to Share IPD: No
Investigators have no reason to disclose participant data but if requested, investigators will share data using the correct necessary steps protecting patient privacy.

REFERENCES:
- [Background] Patel K, Chopra P, Martinez S, Upadhyayula S. Epidural Steroid Injections. 2024 Jun 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470189/ PMID 29262183
- See also: Epidural Steroid Injections — https://www.ncbi.nlm.nih.gov/books/NBK470189/